CLINICAL TRIAL: NCT01027975
Title: Long-term Outcome of Laparoscopic Nissen Fundoplication Compared With Laparoscopic Thal Fundoplication in Children
Brief Title: Comparison of Laparoscopic Nissen Versus Thal Fundoplication in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Mr. Hugh W. Grant , Consultant Paediatric Surgeon, Department of Paediatric Surgery, John Radcliffe Hospital, Oxford, U.K.
Purpose: Treatment
Other Study IDs: RKubiak
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2007-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: laparoscopy; fundoplication; Nissen; Thal; children; operative treatment of gastro-oesophageal reflux disease in children
MeSH Terms: conditions — Gastroesophageal Reflux

INTERVENTIONS:
Procedure: laparoscopic Nissen/laparoscopic Thal

SUMMARY:
Laparoscopic fundoplication is increasingly performed in paediatric surgery. Many types of fundoplication are performed, each has advantages and disadvantages. The Nissen operation is the most frequently performed procedure in the U.K., however it can be associated with post-operative dysphagia. The relative benefits between Nissen and other fundoplication techniques in children are still uncertain.

The aim of our study was to compare the long-term outcomes following laparoscopic Nissen fundoplication with laparoscopic Thal fundoplication in children.

ELIGIBILITY:
Inclusion Criteria:

* Gastro-oesophageal reflux unresponsive to medical treatment, or those who had serious complications (e.g. apnoea, aspiration pneumonia, oesophagitis)

Exclusion Criteria:

* Patients who had previous anti-reflux surgery, previous open abdominal surgery, if parents declined to participate into study

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-07

PRIMARY OUTCOMES:
Recurrence of symptoms sufficiently severe to justify the need for additional revisional surgery (i.e. failure of the original surgery)
Early death following surgery directly related to the fundoplication technique

SECONDARY OUTCOMES:
The resumption of symptoms bad enough to necessitate the re-introduction of anti-reflux medication (but not sufficiently bad to require revisional surgery) i.e. "intention to treat"
Post-operative complications (e.g. post-operative dysphagia)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh W Grant, MD, Study Director — John Radcliffe Hospital, Department of Paediatric Surgery, Oxford,United Kingdom; Rainer Kubiak, MD, Principal Investigator — John Radcliffe Hospital, Department of Paediatric Surgery, Oxford, United Kingdom
Locations (1):
- Department of Paediatric Surgery, John Radcliffe Hospital NHS Trust, Oxford (Headington), Oxford, United Kingdom

REFERENCES:
- [Derived] Kubiak R, Andrews J, Grant HW. Long-term outcome of laparoscopic nissen fundoplication compared with laparoscopic thal fundoplication in children: a prospective, randomized study. Ann Surg. 2011 Jan;253(1):44-9. doi: 10.1097/SLA.0b013e3181fc98a0. PMID 21233605